CLINICAL TRIAL: NCT05760300
Title: A Phase 1 Open-Label, Parallel-Design, Multiple-Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Bulevirtide in Participants With Normal and Impaired Renal Function
Brief Title: A Multiple-Dose Study of Bulevirtide in Participants With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-589-6160; 2022-502054-13-00 (Other: European Medicines Agency)
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis D Infection
MeSH Terms: interventions — bulevirtide; myrcludex-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: BLV 2 mg (Severe RI Group) (Experimental): Participants with severe renal impairment (RI) [estimated glomerular filtration rate (eGFR) ≥ 15 to ≤ 29 mL/min/1.73 m^2] will receive bulevirtide (BLV) 2 mg, administered subcutaneously (SC), once daily (QD), for 6 days.
  Interventions: Drug: Bulevirtide (BLV)
- Group A: BLV 2 mg (Matched Control) (Experimental): Participants with normal renal function (matched control group) [eGFR ≥ 90 mL/min/1.73 m^2] will receive BLV 2 mg, administered SC, QD, for 6 days.
  Interventions: Drug: Bulevirtide (BLV)
- Group B: BLV 10 mg (Severe RI Group) (Experimental): Participants with severe RI [eGFR ≥ 15 to ≤ 29 mL/min/1.73 m^2] will receive BLV 10 mg, administered SC, QD, for 6 days.
  Interventions: Drug: Bulevirtide (BLV)
- Group B: BLV 10 mg (Matched Control) (Experimental): Participants with normal renal function (matched control group) [eGFR ≥ 90 mL/min/1.73 m^2] will receive BLV 10 mg, administered SC, QD, for 6 days.
  Interventions: Drug: Bulevirtide (BLV)

INTERVENTIONS:
Drug: Bulevirtide (BLV) — Administered via subcutaneous (SC) injections
  Other Names: Hepcludex®; Myrcludex B

SUMMARY:
The goals of this study are to compare the amount of study drug, bulevirtide (BLV), that gets into the bloodstream and how long it takes for the body to eliminate it, measure the effect of BLV on bile acids, and evaluate the safety and tolerability of multiple doses of BLV in participants with normal or impaired renal (kidney) function.

ELIGIBILITY:
Key Inclusion Criteria:

All Individuals:

* Body mass index (BMI) of at least ≥ 18.0 kg/m^2 and ≤ 40.0 kg/m^2 at screening.
* No clinically significant abnormalities on electrocardiogram (ECG)
* No known Liver Disease (Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT)) ≤ 3 x upper limit of normal (ULN) at screening.

Individuals with Renal Impairment (RI):

* Have RI classification at screening that has been unchanged during the 90 days prior to study drug dosing.
* Estimated Glomerular Filtration Rate (eGFR) must be the following (using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Inker 2021)) based on serum creatinine as measured at the screening evaluation:

  * Severe RI (Groups A and B): eGFR ≥ 15 to ≤ 29 mL/min/1.73 m^2
  * Moderate RI (Group C): eGFR ≥ 30 to ≤ 59 mL/min/1.73 m^2
  * Mild RI (Group D): eGFR ≥ 60 to ≤ 89 mL/min/1.73 m^2
* Hemoglobin ≥ 9 g/dL at screening.
* Individuals with cardiovascular disease, hypertension, diabetes mellitus, hyperlipidemia, hypothyroidism, osteoporosis, and many others) may be included provided that these diseases/conditions are clinically stable.

Matched Control Individuals:

* Have an eGFR of at least 90 mL/min/1.73 m^2 (using the CKD-EPI equation) based on serum creatinine as measured at screening evaluation.
* Matched for sex, age (± 10 years), and BMI (± 20%, 18.0 ≤ BMI ≤ 40.0 kg/m^2) with the respective participant in the RI group.

Key Exclusion Criteria:

All Individuals:

* Positive human immunodeficiency virus (HIV) test, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody with detectable HCV viral ribonucleic acid (RNA) at screening.
* Have any serious or active medical or psychiatric illness (including depression) that, in the opinion of the investigator, would interfere with participant treatment, assessment, or compliance with the protocol.

Individuals with RI:

* Recent history of reception of any blood or blood products or history of major bleeding within 4 weeks of dosing.
* Positive test for drugs of abuse, including alcohol at screening or admission, with the exception of opioids and tetrahydrocannabinol (THC, marijuana) under prescription and verified by the investigator as for pain management.
* Received treatment with trimethoprim or cimetidine or tenofovir prodrugs (tenofovir disoproxil fumarate (TDF) or tenofovir alafenamide (TAF)) (affects elimination of creatinine) or with competitors of renal tubular excretion (eg, probenecid, chronic high-dose nonsteroidal anti-inflammatory drugs) within 28 days of Day -1.
* Received known nephrotoxic drugs (eg, aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cisplatin, pentamidine, cyclosporine, tacrolimus, herbal remedies (eg, compounds with aristolochic acid)) within 28 days of Day -1.
* Individuals requiring or anticipated to require dialysis within 90 days of study entry.
* Serum albumin concentration <25 g/L.
* Uncontrolled treated/untreated hypertension (defined as a mean of 3 repeated measurements for systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg); current or documented history of repeated clinically significant hypotension or severe episodes of orthostatic hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg).

Matched Control Individuals:

* Have taken any prescription medications or over-the-counter medications, including herbal products, within 28 days prior to start of study drug dosing, with the exception of vitamins

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- United States (9):
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Global Clinical Professionals Research, St. Petersburg, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Massachusetts General Hospital - Renal Associates Clinic, Boston, Massachusetts
  - Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yehong Wang, Renee-Claude Mercier, Wildaliz Nieves, David Pan, Carrie Nielson, SteveTseng, Xu Zhang, Ann Qin, Parag Kumar. Pharmacokinetics, Pharmacodynamics, and Safety of Bulevirtide 2 mg Once Daily for 6 Days in Participants with Severe Renal Impairment and in Matched Control Participants with Normal Renal Function. The Liver Meeting, American Association for the Study of Liver Diseases; November 15-19, 2024; San Diego, CA. Abstract #1194.
- [Background] Yehong Wang, Renee-Claude Mercier, Wildaliz Nieves, Carolina Machado, Steve Tseng, Yuejiao Jiang, Ann Qin, Teckla Akinyi, Parag Kumar, WED-313 Pharmacokinetics, pharmacodynamics, and safety of bulevirtide 10 mg once daily for 6 days in participants with severe renal impairment and in matched control participants with normal renal function, Journal of Hepatology, Volume 82, Supplement 1, 2025, Page S824 (https://doi.org/10.1016/S0168-8278(25)02119-1).
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT05760300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 98 participants were screened. The optional Groups C and D were not initiated and no participants were enrolled in these groups.
Groups:
- Group A: BLV 2 mg (Severe RI Group): Participants with severe renal impairment (RI) [estimated glomerular filtration rate (eGFR) ≥ 15 to ≤ 29 mL/min/1.73 m^2] received bulevirtide (BLV) 2 mg, administered subcutaneously (SC), once daily (QD), for 6 days.
- Group A: BLV 2 mg (Matched Control): Participants with normal renal function (matched control group) [eGFR ≥ 90 mL/min/1.73 m^2] received BLV 2 mg, administered SC, QD, for 6 days.
- Group B: BLV 10 mg (Severe RI Group): Participants with severe RI [eGFR ≥ 15 to ≤ 29 mL/min/1.73 m^2] received BLV 10 mg, administered SC, QD, for 6 days.
- Group B: BLV 10 mg (Matched Control): Participants with normal renal function (matched control group) [eGFR ≥ 90 mL/min/1.73 m^2] received BLV 10 mg, administered SC, QD, for 6 days.
Period: Overall Study
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Started | 10 | 10 | 11 | 10
Completed | 9 | 10 | 10 | 10
Not Completed | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Participant Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug BLV.
Groups:
- Group A: BLV 2 mg (Severe RI Group): Participants with severe RI [eGFR ≥ 15 to ≤ 29 mL/min/1.73 m^2] received BLV 2 mg, administered SC, QD, for 6 days.
- Total: Total of all reporting groups
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control) | Total
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15.1) | 55 (10.6) | 63 (11.1) | 57 (10.6) | 59 (11.9)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 65 years | 6 | 9 | 5 | 8 | 28
  >=65 years | 4 | 1 | 6 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 3 | 14
  Male | 6 | 6 | 8 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 8 | 8 | 31
  Not Hispanic or Latino | 3 | 2 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 4 | 0 | 6
  White | 8 | 10 | 7 | 10 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 11 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter for Bulevirtide (BLV): AUCtau
Description: AUCtau is defined as the area under the concentration versus time curve over the dosing interval at steady state at Day 6.
Time Frame: Day 6: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours postdose
Population: The plasma PK Analysis Set included all enrolled participants who received at least 1 dose of BLV and had at least 1 measurable plasma PK concentration data reported by PK laboratory for the respective analyte. Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours(h)*nanograms per milliliter(ng/mL)
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 6 | 6 | 10 | 10
hours(h)*nanograms per milliliter(ng/mL) | 94.6 (29.8) | 112 (32.6) | 1880 (642) | 1810 (560)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 84.5, 90% CI 2-sided [60.1 to 119] — Parametric (normal theory) analysis of covariance (ANOVA) model appropriate for a parallel design with renal function group as a fixed effect was fitted to the natural log-transformed values of the multiple dose PK parameter under evaluation
Statistical Analysis 2: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 104, 90% CI 2-sided [80.8 to 133] — Parametric (normal theory) ANOVA model appropriate for a parallel design with renal function group as a fixed effect was fitted to the natural log-transformed values of the multiple dose PK parameter under evaluation

2. Primary Outcome: PK Parameter for BLV: Cmax ss
Description: Cmax is defined as the maximum observed concentration of drug at steady state at Day 6.
Time Frame: Day 6: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 9 | 10 | 10 | 10
ng/mL | 15.0 (8.11) | 14.6 (9.35) | 311 (110) | 307 (156)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 106, 90% CI 2-sided [63.6 to 175] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 108, 90% CI 2-sided [77.8 to 151] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: PK Parameter for BLV: AUC0-24
Description: AUC0-24 is defined as the concentration of drug over time between time 0 hour and time 24 hours.
Time Frame: Day 1: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 9 | 9 | 10 | 8
h*ng/mL | 46.5 (13.3) | 53.4 (6.77) | 843 (480) | 876 (458)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 83.8, 90% CI 2-sided [67.4 to 104] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 100, 90% CI 2-sided [56.2 to 179] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: PK Parameter for BLV: Cmax
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Day 1: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours postdose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
ng/mL | 12.3 (4.91) | 13.1 (6.49) | 121 (86.2) | 146 (83.9)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 96.5, 90% CI 2-sided [65.1 to 143] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Test type: Other; Geometric Least-squares Mean Ratio = 77.8, 90% CI 2-sided [42.7 to 142] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: PK Parameter for BLV: Tmax
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Day 1: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours postdose; Day 6: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, and 48 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
h
  Tmax (Day 1) | 1.00 [1.00 to 2.00] | 1.00 [0.500 to 2.00] | 4.00 [1.50 to 6.00] | 4.00 [1.50 to 9.00]
  Tmax (Day 6): number analyzed (Participants) | 9 | 10 | 10 | 10
  Tmax (Day 6) | 1.00 [1.00 to 3.00] | 1.50 [1.00 to 6.00] | 3.00 [2.00 to 4.03] | 3.00 [3.00 to 6.00]

6. Secondary Outcome: PK Parameter for BLV: t1/2
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
h
  t1/2 (Day 1): number analyzed (Participants) | 7 | 8 | 10 | 8
  t1/2 (Day 1) | 2.47 [1.32 to 4.34] | 3.95 [1.20 to 6.66] | 2.86 [1.44 to 14.5] | 3.03 [1.53 to 8.23]
  t1/2 (Day 6): number analyzed (Participants) | 9 | 7 | 10 | 10
  t1/2 (Day 6) | 3.98 [2.84 to 8.72] | 4.60 [2.31 to 7.87] | 2.79 [1.46 to 7.47] | 2.75 [1.44 to 3.78]

7. Secondary Outcome: PK Parameter for BLV: CLss/F
Description: CLss/F is defined as the apparent clearance at steady state at Day 6. CLss/F = Dose/AUCtau, where "Dose" is the dose of the drug per interval.
Time Frame: Day 6: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, and 48 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: milliliters per hour (mL/h)
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 9 | 7 | 10 | 10
milliliters per hour (mL/h) | 29.9 (13.4) | 19.1 (7.54) | 5.80 (1.69) | 6.09 (2.22)

8. Secondary Outcome: PK Parameter for BLV: Vss/F
Description: Vss/F is defined as the apparent volume of distribution at steady state at Day 6.
Time Frame: Day 6: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, and 48 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 9 | 7 | 10 | 10
mL | 222 (175) | 121 (69.4) | 24.4 (10.7) | 25.0 (14.2)

9. Secondary Outcome: Pharmacodynamic (PD) Parameter for Total Bile Acids (BA): Cmax
Description: The PD effect of BLV was evaluated on plasma BA in participants with RI compared to matched control participants with normal renal function. Cmax is defined as the maximum observed concentration of total BA. The plasma bile acid panel includes 15 individual bile acids, and total BA is the sum of these 15 components.
Time Frame: as for outcome 5
Population: The plasma PD Biomarker Analysis Set included all enrolled participants who received at least 1 dose of study drug BLV and had at least 1 measurable plasma PD concentration value reported for each respective analyte. Participants in the PD Biomarker Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/L)
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
micromoles per liter (µmol/L)
  Cmax (Day 1) | 13.5 (8.58) | 8.54 (7.02) | 110 (50.6) | 121 (53.6)
  Cmax (Day 6): number analyzed (Participants) | 9 | 10 | 10 | 10
  Cmax (Day 6) | 48.1 (35.4) | 58.2 (24.5) | 168 (83.4) | 207 (52.1)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Day 1; Test type: Other; Geometric Least-squares Mean Ratio = 160, 90% CI 2-sided [97.2 to 263] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Day 6; Test type: Other; Geometric Least-squares Mean Ratio = 65.9, 90% CI 2-sided [35.0 to 124] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Day 1; Test type: Other; Geometric Least-squares Mean Ratio = 86.7, 90% CI 2-sided [53.3 to 141] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Day 6; Test type: Other; Geometric Least-squares Mean Ratio = 72.6, 90% CI 2-sided [50.4 to 105] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: PD Parameter for Total BA: AUC0-24
Description: The PD effect of BLV was evaluated on plasma BA in participants with RI compared to matched control participants with normal renal function. AUC0-24 is defined as the concentration of total BA over time between time 0 hour and time 24 hours. The plasma bile acid panel includes 15 individual bile acids, and total BA is the sum of these 15 components.
Time Frame: Days 1 and 6: Predose (≤ 30 minutes before dose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours postdose
Population: Participants in the PD Biomarker Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*µmol/L
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
h*µmol/L
  AUC0-24 (Day 1) | 166 (109) | 108 (58.8) | 1290 (613) | 1450 (573)
  AUC0-24 (Day 6): number analyzed (Participants) | 9 | 10 | 10 | 10
  AUC0-24 (Day 6) | 581 (442) | 705 (324) | 2120 (1050) | 2710 (669)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Day 1; Test type: Other; Geometric Least-squares Mean Ratio = 139, 90% CI 2-sided [87.8 to 221] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Day 6; Test type: Other; Geometric Least-squares Mean Ratio = 66.8, 90% CI 2-sided [37.3 to 120] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Day 1; Test type: Other; Geometric Least-squares Mean Ratio = 85.7, 90% CI 2-sided [54.5 to 135] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Day 6; Test type: Other; Geometric Least-squares Mean Ratio = 70.3, 90% CI 2-sided [49.4 to 100] — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: PD Parameter for Total BA: NetAUC
Description: The PD effect of BLV was evaluated on plasma BA in participants with RI compared to matched control participants with normal renal function. NetAUC is defined as positive portion of area under the baseline-adjusted biomarker concentration versus time curve over the dosing interval. The plasma bile acid panel includes 15 individual bile acids, and total BA is the sum of these 15 components.
Time Frame: as for outcome 5
Population: Participants in the PD Biomarker Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*µmol/L
Groups:
- Group B: BLV 10 mg (Matched Control): Participants with normal renal function (matched control group) [eGFR ≥ 90 mL/min/1.73 m^2] received BLV 10 mg, administered SC, QD, for 6 days.ays.
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
h*µmol/L
  NetAUC (Day 1) | 54.9 (40.4) | 66.1 (57.6) | 1240 (598) | 1400 (572)
  NetAUC (Day 6): number analyzed (Participants) | 9 | 10 | 10 | 10
  NetAUC (Day 6) | 496 (433) | 662 (330) | 2060 (1020) | 2660 (666)
Statistical Analysis 1: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Day 1; Test type: Other; Geometric Least-squares Mean Ratio = 84.2, 90% CI 2-sided [32.7 to 217] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group A: BLV 2 mg (Severe RI Group) vs Group A: BLV 2 mg (Matched Control); Day 6; Test type: Other; Geometric Least-squares Mean Ratio = 58.0, 90% CI 2-sided [30.1 to 112] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Day 1; Test type: Other; Geometric Least-squares Mean Ratio = 85.6, 90% CI 2-sided [54.1 to 135] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Group B: BLV 10 mg (Severe RI Group) vs Group B: BLV 10 mg (Matched Control); Day 6; Test type: Other; Geometric Least-squares Mean Ratio = 69.6, 90% CI 2-sided [48.9 to 99.2] — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or if the AE onset date was the same as the date of study drug start date then the AE onset time must have been on or after the study drug start time. If the AE onset time was missing when the start dates was the same, the AE was considered treatment emergent.and/or any AEs leading to premature discontinuation of study drug.
Time Frame: Up to 36 days
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug BLV.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
percentage of participants | 40.0 | 20.0 | 27.3 | 30.0

13. Secondary Outcome: Percentage of Participants Experiencing Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was any value that was outside the reference range at any time post baseline up to and including the date of last study drug dose plus 30 days. Grading categories are determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening; Grade 5: Death. Participants with at least a 1 grade increased from baseline for an individual laboratory test where the maximum post baseline laboratory abnormality was grade 1 or higher and grade 3 or higher were reported. The maximum post baseline toxicity grade across all tests for an individual participant was used in analysis.
Time Frame: Up to 36 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Group A: BLV 2 mg (Severe RI Group): PParticipants with severe RI [eGFR ≥ 15 to ≤ 29 mL/min/1.73 m^2] received BLV 2 mg, administered SC, QD, for 6 days.
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
Number analyzed (Participants) | 10 | 10 | 11 | 10
percentage of participants
  Grade 1 or Higher | 100 | 90.0 | 100 | 90.0
  Grade 3 or Higher | 50.0 | 0 | 45.5 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 420 days; Adverse Events: Up to 36 days
Description: All-Cause Mortality: The All Enrolled Analysis Set included all participants who received a study participant identification (ID) number in the study after screening.
  Adverse Events: The Safety Analysis Set included all participants who took at least 1 dose of study drug BLV.
Arm/Group | Group A: BLV 2 mg (Severe RI Group) | Group A: BLV 2 mg (Matched Control) | Group B: BLV 10 mg (Severe RI Group) | Group B: BLV 10 mg (Matched Control)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 2/10 | 2/11 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: BLV 2 mg (Severe RI Group) (N=10) | Group A: BLV 2 mg (Matched Control) (N=10) | Group B: BLV 10 mg (Severe RI Group) (N=11) | Group B: BLV 10 mg (Matched Control) (N=10)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: BLV 2 mg (Severe RI Group) (N=10) | Group A: BLV 2 mg (Matched Control) (N=10) | Group B: BLV 10 mg (Severe RI Group) (N=11) | Group B: BLV 10 mg (Matched Control) (N=10)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT05760300/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT05760300/SAP_001.pdf